CLINICAL TRIAL: NCT02463305
Title: Therapeutic Modulation of the Intestinal Creatine Kinase System in Inflammatory Bowel Disease (IBD)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: inability to enroll
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-3054; UL1TR001082 (NIH)
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, ulcerative; Inflammatory bowel diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Creatine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment arm (Experimental): 6 patients with mild-moderate ulcerative colitis treated with creatine monohydrate 21 grams per day in three divided doses taken with water for 8 weeks.
  Interventions: Drug: Creatine monohydrate
- Placebo arm (Placebo Comparator): 6 patients with mild-moderate ulcerative colitis treated with placebo (matching creatine monohydrate) 21 grams per day in three divided doses taken with water for 8 weeks.
  Interventions: Other: Placebo
- Optional Open-Label Treatment arm (Experimental): Up to 6 patients, who were randomized to the placebo arm, will be given the option to continue with open-label creatine monohydrate treatment at 21 grams per day in three divided doses, taken with water, for 8 weeks. Only non-invasive testing will be performed.
  Interventions: Drug: Creatine monohydrate

INTERVENTIONS:
Drug: Creatine monohydrate — 21 grams creatine monohydrate total per day
  Arms: Optional Open-Label Treatment arm; Treatment arm
Other: Placebo — 7 grams of dextrose dissolved in 500mL water, taken three times daily
  Other Names: Dextrose
  Arms: Placebo arm

SUMMARY:
This study plans to learn more about the effects that creatine monohydrate has on disease activity in ulcerative colitis. Creatine is a substance that is naturally produced by the body and is found in foods, such as meat and fish. Creatine helps to provide energy to some body tissues, such as the colon. In the colon, this energy allows cells to form a tight barrier between molecules in digested food and bacteria and the body's infection-fighting cells within the colon underneath this barrier. If the barrier becomes "leaky" molecules may pass through and lead to inflammation. This "leakiness" may contribute to the colon inflammation seen in ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18-70 years old with mild- to moderately-active UC that extends at least 15 cm proximal to the anal verge (i.e. not proctitis) as defined by a Mayo Score of 3-10, with an endoscopic subscore ≥ 1.
* Allowed concomitant medications will include mesalamine compounds if used for at least 8 weeks and at a stable dose for at least 4 weeks, as well as thiopurines (azathioprine, 6-mercaptopurine) if used at a stable dose for at least 3 months.

Exclusion Criteria:

* Abnormal baseline laboratory tests:

  * Albumin < 3.0 g/dL
  * ALT, AST, total bilirubin, or alkaline phosphatase > 1.5 x ULN
  * Potassium < 3.0 mmol/L or > 5.5 mmol/L
  * Creatinine or cystatin C > ULN
  * WBC ≤ 3000
  * Platelets ≤ 105
  * Hemoglobin ≤ 10g/dL
  * Positive stool test for Clostridium difficile, ova and parasites, or routine stool culture
* Pregnancy (as confirmed by urine pregnancy test at study outset), stated desire to become pregnant during the study period, or refusal/inability to use effective methods of contraception during the study period.
* Concomitant major comorbidities (renal, hepatic, cardiac, pulmonary or malignancy) to include any medical conditions requiring therapeutic anti-coagulation or anti-platelet therapy.
* Diagnosis of severe UC (Mayo Score > 10)
* Evidence or history of toxic megacolon
* Patients who received anti-TNF agents within 3 months of screening, or who used oral or rectal corticosteroids within 4 weeks of screening will be excluded.
* Use of over-the-counter herbal or dietary supplements (excluding vitamin and minerals) two weeks prior to or during the study period.
* Use of known nephrotoxic medications (including non-steroidal anti-inflammatory drugs (NSAIDs), cyclosporin A, tacrolimus, aminoglycoside antibiotics, diuretics, angiotensin converting enzyme (ACE) inhibitors, or angiotensin receptor blockers) 2 weeks prior to or during the study period
* Prior surgical bowel resections (excluding appendectomy)
* Local or systemic complications or other pathological states requiring therapy with corticosteroids and/or immunosuppressive agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Improvement in endoscopic assessment of mucosal inflammation in ulcerative colitis. | 8 weeks
  As defined by the Mayo endoscopic score for ulcerative colitis.

SECONDARY OUTCOMES:
Clinical response in ulcerative colitis disease activity. | 8 weeks
  As defined by the Mayo composite score for ulcerative colitis.
Intestinal permeability | 8 weeks
  As measured by urinary saccharide excretion
Patient symptom severity | 8 weeks
  As measured by inflammatory bowel disease questionnaire (IBDQ), simple Crohn's and colitis activity index (SCCAI), and Mayo composite scores.
Colonic inflammation | 8 weeks
  As assessed by fecal calprotectin, CRP, and histologic scoring.
Creatine kinase modulation | 8 weeks
  As assessed by CK transcript and protein in colonic tissue and serum levels.
Clinical remission of ulcerative colitis disease activity. | 8 weeks
  As defined by the Mayo composite score for ulcerative colitis.
Creatine modulation | 8 weeks
  As defined by colonic tissue and serum levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gerich, MD, Principal Investigator — University of Colorado Denver, Division of Gastroenterology
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No